CLINICAL TRIAL: NCT03498599
Title: Improving the Control of Fear: Healthy Adults to Pathological Anxiety
Brief Title: Neuroimaging of Pavlovian Fear Conditioning Processes in Patients With Pathological Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UTfearconditioning
Record Dates: First submitted 2018-02-15; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Post Traumatic Stress Disorder; Anxiety Disorders; Panic Disorder; Social Phobia; Phobia
Keywords: neuroimaging; fear conditioning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Panic Disorder; Phobia, Social; Phobic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novelty facilitated extinction (Experimental): Behavioral intervention. After Pavlovian fear conditioning, the shock is omitted and replaced by a novel, surprising, and neutral auditory tone.
  Interventions: Behavioral: Novelty facilitated extinction
- Standard extinction (Other): The shock is omitted during standard extinction
  Interventions: Behavioral: Standard Extinction

INTERVENTIONS:
Behavioral: Novelty facilitated extinction — In the novelty-facilitated extinction design, the aversive outcome (i.e., mild unpleasant electrical pulse) is omitted and replaced by a low volume auditory tone.
  Arms: Novelty facilitated extinction
Behavioral: Standard Extinction — During standard fear extinction the expected aversive outcome is omitted.
  Arms: Standard extinction

SUMMARY:
The purpose of this study is to use functional magnetic resonance imaging to investigate how the human brain learns to form associations between neutral and emotional stimuli. The study is based on the basic principles of Pavlovian conditioning.

When someone learns that a neutral stimulus (such as the sound of a bell) predicts an unpleasant stimulus (such as a mild electrical shock), the neutral stimulus takes on the properties of an emotional stimulus.

The investigators are interested in the neural processes involved in this learning in people with a clinical anxiety disorder and posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
This study uses functional MRI in people with anxiety and stress-related disorders to evaluate the neural correlates of fear conditioning and extinction. During fear conditioning participants see a picture of a face that predicts a mild electrical shock to the wrist. Participants then return the next day to the scanner for a test of fear expression 24-hours after fear conditioning. The investigators are simultaneously measuring autonomic arousal in the scanner using measures of skin conductance responses (i.e., sweating).

The primary objective of this study is to evaluate different forms of Pavlovian fear extinction in patients who suffer from pathological anxiety. The investigators are interested in the effects of extinction and extinction retention over a delay in regions that are known to show abnormalities in anxiety populations. This includes the amygdala, ventromedial prefrontal cortex, and the hippocampus.

The study is testing behavioral strategies and does not include any pharmacological manipulations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteer aged 18-50 years old
2. Able to understand procedures and agree to participate in the study by giving written informed consent.
3. Speaks fluent English.
4. Not taking illicit drugs.
5. No history of neurological problems.
6. Eligible for MRI, including no metal in the body or body piercings that cannot be removed.

Exclusion Criteria:

1. Current comorbid Axis 1 psychiatric disorder
2. Women who are current pregnant or breastfeeding
3. Lifetime diagnosis of any psychotic disorder, cognitive suicidal ideation, substance abuse or alcohol dependence, hoarding.
4. Medications that act on the central nervous system that interfere with interpretation of the findings (e.g., painkillers, Adderall)
5. Claustrophobia
6. Patients who are unable to comply with procedures or assessments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Changes in functional magnetic resonance imaging (fMRI)-BOLD (blood-oxygen-level dependent) signal in sensory, prefrontal, and limbic regions during a study on the neurobiology of Pavlovian fear conditioning in humans | Only on the day of the experiment
  We are measuring increases in the BOLD signal in response to visual stimuli during a Pavlovian conditioning task in humans.

SECONDARY OUTCOMES:
Skin conductance responses evoked during a Pavlovian fear conditioning task in humans as an index of physiological arousal. | Only on the day of the experiment
  Electrodermal activity collected from the hand that measures increases in sweating, taken as an indicator of Pavlovian fear conditioning

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH Data Archive
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Less than 6 months after data is collected.
Access Criteria: We will upload data to the NIMH Data Archive and data will be accessible per their policy.